CLINICAL TRIAL: NCT04291222
Title: Feasibility, Efficacy and Safety of IBS ® for Implantaiton in the PDA in Duct-dependent Cyanotic CHD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Lifetech Scientific (Shenzhen) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IBS-AngelV1.0
Record Dates: First submitted 2020-02-28; First posted 2020-03-02 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Patent Ductus Arteriosus; Duct-dependent Cyanotic Congenital Heart Disease
MeSH Terms: conditions — Ductus Arteriosus, Patent

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IBS implantation (Experimental): Implantation of IBS in PDA in duct-dependent cyanotic CHD
  Interventions: Device: Iron biocorrodable coronary scaffold system

INTERVENTIONS:
Device: Iron biocorrodable coronary scaffold system — Implantation of Iron biocorrodable coronary scaffold system

SUMMARY:
This is a pilot study on feasibility, efficacy and safety of IBS ® for implantation in the PDA in duct-dependent cyanotic CHD, and its objective is to investigate the feasibility, safety and efficacy of iron resorbable stent implantation in the PDA as initial palliation of cyanotic CHD with duct-dependent PBF.

DETAILED DESCRIPTION:
Study type: Interventional, prospective, single arm, investigator initiated Study population: 10 patients Primary purpose: Treatment Follow up: Review at 1 month and thereafter 3 monthly (clinical examination and echocardiography for stent patency, SaO2 measurement. Serum Iron and Ferritin levels will be measured before procedure and at follow ups. From 6 months onwards the patients will be assessed for the need of repeat catheterization with a view of surgery or for continued observation.

Study endpoints: 9 months post implant or the following: 1)Patients are subjected for surgical repair of CHD; 2)Death before surgical repair; 3)Unplanned re-intervention with additional stenting procedure.

ELIGIBILITY:
Inclusion Criteria:

* Weight >3.0 kg
* Age <3 months
* Patients with uncomplicated PDA morphology (the PDA is not tortuous i.e. relatively straight

Exclusion Criteria:

* Weight <3 kg, age >3 months
* Angiographic criteria-tortuous PDA
* Family history of diseases related to iron overload or iron disorder e.g. hereditary hemochromatosis
* Other severe congenital anomalies with life expectancy <12 months

Max Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2018-12-11 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Number of participants for surgical repair of CHD | 9 months
  Patients are subjected for surgical repair of CHD
Number of Unplanned re-intervention | 9 months
  Unplanned re-intervention with additional stenting procedure
Death | 9 months
  Death before surgical repair

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Jantung Negara, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided